CLINICAL TRIAL: NCT06847412
Title: Comparative Study of Escalating PEEP (Positive End Expiratory Pressure) vs. Lung Recruitment by Sustained Inflation Strategies for Managing Hypoxemia in COPD Patients Undergoing Video-Assisted Thoracoscopic Surgery (VATS)
Brief Title: The Effectiveness of Two Distinct Ventilation Strategies Escalating Positive End Expiratory Pressure (PEEP) and Lung Recruitment Maneuvers in Improving Oxygenation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MS 40/2025
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: Hypoxemia; COPD
MeSH Terms: conditions — Hypoxia; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (A): Escalating PEEP (Active Comparator): This group will undergo VATS & one hypoxemia started PEEP is typically increased in 2-3 cm H₂O increments while monitoring the patient's response (oxygenation, hemodynamics, and lung compliance).
  Interventions: Device: Escalating PEEP
- Group (B): Lung recruitment by Sustained inflation (Active Comparator): A sustained inflation:
  Set the ventilator to CPAP mode and increase the pressure to 30 cm H2O for 30 s.
  Interventions: Device: Sustained inflation

INTERVENTIONS:
Device: Escalating PEEP — Typically, an initial PEEP of 5 cm H₂O, then PEEP is increased in 2-3 cm H₂O increments while monitoring the patient's response (oxygenation, hemodynamics, and lung compliance).
  Arms: Group (A): Escalating PEEP
Device: Sustained inflation — Set the ventilator to CPAP mode and increase the pressure to 30 cm H2O for 30 s.
  Arms: Group (B): Lung recruitment by Sustained inflation

SUMMARY:
This study evaluates and compares the effectiveness of two distinct ventilation strategies-escalating PEEP and lung recruitment maneuvers-in improving oxygenation (i.e., managing hypoxemia) in COPD patients undergoing VATS.

DETAILED DESCRIPTION:
A) Preoperative settings :

* Written informed consent will be obtained from all participants prior to the study.
* Pre-operative optimisation of patients include cessation of smoking, improvement of pulmonary functions using bronchodilators and steroids, pre-operative chest physiotherapy and training of patient with lung expansion manuoevers. Reversible components of COPD such as bronchospasm, infections, and pulmonary oedema should be actively looked for and treated aggressively 9.
* Detection of severity of COPD by using The Global Initiative for Chronic Obstructive Lung Disease (GOLD) system categorizes airflow limitation into stages. In patients with FEV₁/FVC <0.7:

  * GOLD 1 - mild: FEV₁ ≥80% predicted
  * GOLD 2 - moderate: 50% ≤ FEV₁ <80% predicted
  * GOLD 3 - severe: 30% ≤ FEV₁ <50% predicted
  * GOLD 4 - very severe: FEV₁ <30% predicted 10.
* Preoperative assessment evaluates lung mechanics, parenchymal function, and cardiopulmonary reserve to determine a patient's suitability for surgery. Lung mechanics, including forced expiratory volume in 1 second (FEV1), maximum voluntary ventilation, forced vital capacity, and residual volume/total lung capacity (RV/TLC) ratio, provide insights into respiratory function. An FEV1 greater than 60% indicates potential tolerance for anatomic lobe resection. An FEV1 of less than 30% suggests postoperative ventilator or supplemental oxygen dependence. In FEV1s less than 60%, a ventilation-perfusion scan (VQ scan) may calculate a postoperative FEV1, with values above 35% (and up to 40%), suggesting adequate postoperative pulmonary reserve. DLCO, measuring gas diffusion, ideally exceeds 40% for surgery. Cardiopulmonary exercise testing assesses overall reserve, with a maximum rate of oxygen (O2) your body can use during exercise (VO2) greater than 10 mL/min/kg, indicating suitability for surgery 2.
* Preoperative assessment for VATS also involves evaluating blood counts for indications of polycythemia or infection. Chest x-rays and CT scans provide anatomical details for surgical planning. Arterial blood gases identify patients at risk for postoperative complications; a partial pressure of carbon dioxide (CO2) more than 50 mm Hg or a partial pressure of O2 less than 60 mm Hg indicates vulnerability 2.

B) Intraoperative settings:

Electrocardiogram (ECG), non-invasive blood pressure (NIBP), pulse oximeter (SpO2) will be applied, and baseline readings will be taken before induction.

Anaesthesia will be induced after a period of preoxygenation with 100% oxygen for 2-3 minutes with intravenous injection of fentanyl 2 µg/kg, propofol 2 mg/kg and a muscle relaxant (Atracurium) 0.5 mg/kg after loss of patient consciousness. Lung isolation is achieved using a double-lumen endotracheal tube, Fiberoptic bronchoscopy is typically used to guide and confirm the placement and positioning of the tube 11.

Patients often requires the placement of invasive monitoring devices, such as invasive blood pressure (IBP) lines and central venous lines (CVL).

Anaesthesia will be maintained by 1-2 % of isoflurane in 50% oxygen/air mixture according to oxygen state and 0.1 mg/kg atracurium, ventilation parameters that maintain normocapnia (CO2 between 35- 40 mmHg). Fluids as crystalloids used by a fluid chart for the deficit and maintenance as needed.

The surgery typically begins with the patient positioned in a full lateral decubitus posture tailored to the side of the operation or in a supine position with appropriate support to access the chest.

Ventilatory setting:

Typically, an initial PEEP of 5 cm H₂O is used in all patients,

Group A:

PEEP is typically increased in 2-3 cm H₂O increments while monitoring the patient's response (oxygenation, hemodynamics, and lung compliance).

Group B:

A sustained inflation:

Set the ventilator to CPAP mode and increase the pressure to 30 cm H2O for 30 s.

C) Postoperative settings:

Follow up patients in recovery room whether transferred to ICU or to Ward, data will be recorded at the following times 1 h, 2 h, 6 h, 12 h, and 24 h. Both groups will be compared to each other according to the following variables:

* Hypoxemia
* The Need for mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years and </=60 years.
* Both sex.
* Patients American Society of Anesthesiologists Physical Status (ASA) Il to IIl.
* A written, valid, and informed consent
* Mild to moderate COPD patients
* BMI less than 4

Exclusion Criteria:

* Patient refusal.
* Pregnancy
* VATS procedure converted to open thoracotomy
* Patients have other lung diseases
* Patients ASA more than lll
* Patients with cardiac diseases affecting systolic & diastolic functions

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-07-27 (Estimated); Study Completion 2025-07-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of ICU admission | 6 months
  The incidence of post-operative patients requiring ICU admission

SECONDARY OUTCOMES:
Incidence of pulmonary complications | 6 months
  Intraoperative Hemodynamic instability, hypoxemia & Hypercapnia Post operative Needs of mechanical ventilation. Post operative pulmonary complications.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Nagah AL Shaer, Professor, Study Chair — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All dana will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before 1/2026
Access Criteria: Free